CLINICAL TRIAL: NCT06786949
Title: Night-shift Work and Breast Cancer
Acronym: BC-NSW-02/2023
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: BC-NSW-02/2023; PNRR-MAD-2022-12376823 (Other Grant/Funding Number: NexTGeneration EU)
Record Dates: First submitted 2025-01-02; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Risk Factors
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subgroup 1: For the analysis of possible risk factors for breast cancer (secondary objective 1), a nested case-control study will be conducted on a subpopulation of the health worker cohort: 100 cases will be selected from the health workers in the cohort who have been diagnosed with breast cancer; 3 healthy controls will be selected for each case (300 total) and will be matched to the cases based on center, age, and period of first employment
  Interventions: Other: Questionnaire
- Subgroup 2: For the measurement of biomarkers of aging whose expression might be associated with night shifts (secondary objective 2), 200 health care workers who have been exposed to at least 6 night shifts per month in the past 6 months and 200 unexposed health care workers, plus 50 other health care workers in each group to prevent possible nonadherence to the study, will be randomly selected from the cohort of health care workers currently still in service.
  Interventions: Diagnostic Test: Blood samples for biomarker measurement

INTERVENTIONS:
Other: Questionnaire — All cases and controls will be contacted by telephone or e-mail and invited to participate in the study. Female workers who decide to join the study will be asked to go to their company's occupational health clinic where they will undergo administration of a questionnaire to investigate possible known and unknown risk factors for breast cancer
  Groups: Subgroup 1
Diagnostic Test: Blood samples for biomarker measurement — Women who give consent to undergo this phase of the study will be called back to the center and will be asked to provide a blood sample
  Groups: Subgroup 2

SUMMARY:
Scientific evidence established about the effects of night work on health both in the short term (insomnia, excessive sleepiness, difficulty concentrating or lack of energy) and in the long term (moderately high risk of developing cardiovascular disease, type 2 diabetes, depression, cancer). In light of the scientific evidence, the IARC (International Agency for Research on Cancer) has listed night work as a probable human carcinogen (Group 2). With respect to current knowledge, the present study could provide valuable help in understanding the mechanisms by which circadian rhythm alteration acts at the genetic level in terms of promoting oncogenesis. Furthermore, by studying its association with other risk factors, understand whether there is a pattern of women more susceptible to its oncopromoting action.

DETAILED DESCRIPTION:
Certain bodily functions, such as wakefulness and sleep, regulation of blood pressure and body temperature, the immune system, gene expression, and secretion of hormones--think of cortisol, for example--follow variations that are stably repeated every 24 to 25 hours. The biological clock that marks this cyclical rhythm is represented by neurons in the suprachiasmatic nucleus of the hypothalamus. Of the circadian system, three components should be considered: (a) the input pathways that transmit signals to synchronize the endogenous central clock with the external environment, (b) the central clock generates rhythms, and (c) the output pathways that transmit the signal from the central clock to other regulatory systems in the brain and body. The most powerful regulator of the input pathways is light, which-as is well known-is captured by the five retinal photoreceptors, including the intrinsically photosensitive retinal ganglion cells [ipRGCs], which, through the production of melanopsin, transmit the signal to the central circadian clock. Such physiological mechanisms, which have remained unperturbed for thousands of years, have been disrupted by the spread of artificial lighting, which, inevitably, alters the natural synchronization of the internal clock with sunlight.

The effects that this misalignment produces are clearly visible in night workers who frequently have to expose themselves to light at "atypical" hours. In this sense, in fact, according to current legislation (see Art. 1, Legislative Decree No. 66 of April 8, 2003, implementing Directives 93/104/EC and 2000/34/EC, concerning certain aspects of the organization of working time), a night worker is defined as anyone who works for a period of at least seven consecutive hours including the interval between midnight and 5 a.m. It follows with palpable evidence that there is an increased risk that, under night work conditions, the alteration of the sleep-wake rhythm may take on a chronic character. In this regard, scientific evidence about the effects of night work on short-term health is well established: such as insomnia, excessive sleepiness, difficulty in concentration or lack of energy. While there is also scientific evidence that some repercussions may also occur in the long term. This is, in that case, the moderately high risk of developing cardiovascular disease, type 2 diabetes, depression, and, not least, cancer. Indeed, in 2007, in light of scientific evidence, the IARC (International Agency for Research on Cancer) listed night work as a probable human carcinogen (Group 2). Breast cancer generally represents the second most frequent neoplastic disease in women. The incidence of new cases worldwide in 2017 was estimated to be 1.9 million, higher in industrialized countries. From a pathogenetic point of view, the association between night shift work and breast cancer is highly plausible.

ELIGIBILITY:
Inclusion Criteria:

* Health workers with any type of contract and qualification (doctors, nurses, OSS) in service at IRCSS AOUBO and AOU "G. Martino" of Messina for at least six months between 1.1.2000 and 31.12.2021
* Age between 20 and 70 years at the start of study follow-up (6 months after recruitment or 1.1.2000)
* Female gender
* For secondary objective 2 of the study only, women exposed to night work must have worked at least 6 night shifts per month in the past six months

Exclusion Criteria:

* Women found to be positive for BRCA1 and BRCA2 genetic mutation (BRCA1 and 2 mutations are searched for by geneticists in sick women for whom there is a consistent suspicion of mutation)
* Women with prior history of breast cancer at the time of recruitment or within six months thereafter.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Health care workers with an employment relationship at IRCCS AOUBO Policlinico di S. Orsola and AOU "G. Martino" of Messina undergoing health surveillance, aged between 20 and 70 years at the time of recruitment (from January 1, 2000 until December 31, 2021).
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Estimate the relationship between exposure to night work and breast cancer incidence | through study completion, an average of 1 year
  The primary objective of the study is to estimate the relationship between exposure to night work and incidence of breast cancer in a cohort of female health care workers who have been in service at IRCCS AOUBO Policlinico di S. Orsola and Azienda Ospedaliero- Universitaria "G. Martino" in Messina.

SECONDARY OUTCOMES:
Identify by case-control analysis which risk factors are associated with the development of breast cancer | Six months from the start of follow-up
  identify by case-control analysis which risk factors are associated with the development of breast cancer and evaluate their effect on the relationship between exposure to night work and breast cancer occurrence among female health workers in the selected cohort
Determine whether epigenetic alterations are more prevalent in the genome of women exposed to night work | At enrollment in the study
  Determine whether epigenetic alterations attributable to the effect of altered sleep-wake rhythm are more present in the genome of women exposed to night work than in women not exposed to night work.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Violante, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- Italy (2):
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, U.O. Medicina del Lavoro, Bologna
  - AOU G. Martino Messina U.O.S.D. Medicina del Lavoro, Messina